CLINICAL TRIAL: NCT01333371
Title: Are Volar Locking Plates a Cost Effective Strategy for the Treatment of Distal Radius Fractures in Patients <65 Years of Age?
Brief Title: Assessing Volar Locking Plates in Patients Under 65 With a Distal Radius Fracture
Acronym: DRF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hand and Upper Limb Clinic, Canada (Network)
Collaborators: Canadian Orthopaedic Foundation (Other)
Responsible Party: Dr. Ruby Grewal, Hand and Upper limb Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HULC drf-Volar Plate; 17545 (Other Grant/Funding Number: Canadian Orthopedic Foundation Department of Surgery Internal Research Fund)
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Distal Radius Fracture
Keywords: Distal Radius; Volar locked plating; Cost Effectiveness; Randomization; Outcomes
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- closed reduction with percutaneous k-wire fixation and casted (Active Comparator)
  Interventions: Procedure: Surgical Repair of Distal Radius Fracture
- open reduction internal fixation with a volar locked plate (Active Comparator)
  Interventions: Procedure: Surgical Repair of Distal Radius Fracture

INTERVENTIONS:
Procedure: Surgical Repair of Distal Radius Fracture — 2 surgical methods to treat Distal Radius Fracture

SUMMARY:
Patients will be randomized to volar plating with early ROM versus closed reduction with K-wires and 6 weeks of cast immobilization to determine if there is any advantage to volar plating in this subgroup of patients with distal radius fractures.

DETAILED DESCRIPTION:
This study has been designed as a prospective randomized controlled trial examining the cost effectiveness of treating distal radius fractures with open reduction and internal fixation with a volar locking plate (VLP) to closed reduction and k-wire fixation (K-Wires). All patients aged < 65 years with an isolated distal radius fracture (extra-articular or simple intra-articular, AO type A or C1) requiring operative fixation will be included in this study. Patients who have underlying osteoporosis, other injuries or complex intra-articular fractures will be excluded from this study.

Once eligibility is determined, patients will be randomized to one of two treatment arms. They will be treated with either a closed reduction with percutaneous k-wire fixation and 6 weeks of cast immobilization (K-wire) or open reduction internal fixation with a volar locked plate and early range of motion (beginning at 10-14 days) (VLP). All patients will undergo a standardized pre-operative evaluation. This will include classification of their fracture (based on the AO classification), a baseline PRWE and DASH score, a measure of their general health (SF-12) and a general health utility questionnaire (EQ-5d). Patients will be required to report the details of their occupational physical demands and the number of work days missed due to injury.

Patient testing will be incorporated into scheduled clinic visits. Data will be collected at the initial assessment, 2 weeks post-operatively, and then at 6 weeks, 12 weeks, 6 months and 12 months after the fracture. At each visit, AP and lateral wrist radiographs will also be obtained. The investigators will then examine the outcomes of each group based on range of motion, grip strength, and standardized patient rated pain and disability scores (PRWE and DASH). In order to capture differences between the 2 groups in the early phases of recovery - the investigators will administer 2 additional assessments at 4 and 9 weeks by either phone or email. These telephone assessments will include an assessment of patient rated pain and disability (DASH, PRWE) and patients will be asked to provide details on whether they have returned to work or their usual activities.

The primary outcome, patient rated pain and disability, will be quantified with the Patient Rated Wrist Evaluation (PRWE) a tool which has been shown to be valid, reliable and highly responsive in the distal radius fracture population. Secondary outcomes will include range of motion, strength, Disabilities of Arm Shoulder and Hand Score (DASH) and time to return to work. The cost analysis will include both direct and indirect costs, and will include: OR time, anesthesia time, surgeon fees, cost of outpatient visits, equipment costs (volar locked plates and k-wires), x-rays, casting, splints, number of work days missed and work disability costs. The investigators will also use the health utility score (EQ-5d) to determine the cost per quality adjusted life year (QALY) associated with each intervention.

Based on our sample size calculations, the investigators will need 28 patients in each treatment arm (power 80%, p = 0.05). Allowing for a 10-15% drop-out rate, 64 patients are required for enrollment. The secondary outcomes will include ROM, grip strength, union rate, mean time to union (weeks) and DASH score.

ELIGIBILITY:
Inclusion Criteria:

* Distal radius fracture - AO type A or C1
* Skeletally mature
* Age 18-65 years old
* Isolated injury

Exclusion Criteria:

* AO Type B or C2,3
* Other injuries involving affected or unaffected arm
* Skeletally immature

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Patient Rated Wrist Evaluation | Prior to randomization and at 3, 6, and 12 months following randomization
  Questionnaire administered to assess subjective levels of pain and function

SECONDARY OUTCOMES:
Objective measures | 3, 6, and 12 months following surgery
  ROM, Strength and Dexterity will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Ruby Grewal, MD, FRCSC, Principal Investigator — Hand and Upper Limb Clinic, St. Joseph's Health Care
Locations (1):
- Hand and Upper Limb Clinic, St Joseph's Health Care, London, Ontario, Canada